CLINICAL TRIAL: NCT06193785
Title: Evaluation of Hypnosis Practice During a Semi-invasive and Painful Medical Examination in Neurology: the Electromyogram
Acronym: HYPNOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHPAU2023/02
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Patients Requiring Electromyogram
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Prospective therapeutic study comparing two groups, open, quasi-randomised, single-centre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): hypnosis realised by expert practitioner during electromyogram realisation
  Interventions: Other: Hypnosis
- control (No Intervention): standard electromyogram realisation

INTERVENTIONS:
Other: Hypnosis — hypnosis realised by expert practitioner, before and during the electromyogram procedure
  Arms: Hypnosis

SUMMARY:
Electromyogram is a current exam usually in neurological practices use for study peripheral nervous system. This is a semi-invasive examination causing pain. The aim of the study is to evaluate hypnosis practice in patients during an electromyogram. The investigator will evaluate pain with quantitative and qualitative evaluation in two groups with and without hypnosis in an open, quasi-randomised prospective therapeutic study in Pau hospital centre

DETAILED DESCRIPTION:
Electromyogram is frequently use in neurological practices for neuropathies detection or others peripheral nervous system affection. There is two parts during this examination. The first is called sensory and motor nervous conduction study. It consists to apply cutaneous electrodes wich send electric current on arms and legs. The second is the detection with use needles in several muscles of the four limbs with muscle contraction. So, electromyogram is long (sometimes up to one hour) and painful assessment.

Hypnosis is an old not invasive easy practice using in some medical conditions like fibroscopy, anesthesia, surgery. The mechanisms are unclear but this is an effective practice particularly in pain management. Hypnosis in neurological examinations remains unusual. Only two studies report use of hypnosis during electromyogram. The first in 2009 is a randomised suty. On 26 patients, they study hypnosis impact on anxiety and pain. The conclusion is significant efficacity of hypnosis on pain during electromyogram with pain decrease of 31% compared with control group. The second is a French study with only poster. There was no significant difference between hypnosis group and control group during electromyogram for pain. But, there was significant difference for anxiety item. These two studies shown opposite results.

In this study, the sponsor propose to evaluate hypnosis during electromyogram. The main criteria is quantitative pain evaluation. A neurologist doctor will do electromyogram and specialized nurse will do hypnosis. This is a prospective open, quasi-randomised study with two groups of patients. One with hypnosis realised by expert practitioner during electromyogram realisation. One group without hypnosis. The investigator will note pain during examination with standardised quantitative (primary outcome) and qualitative (secondary outcome) evaluation. The investigator will use visual Analog Scale and Saint-Antoine Pain Questionary (QDSA) but also Beck Anxiety Inventory for psychological effect. The duration of study is one year in single centre. The Pau Hospital hope validate this practice of hypnosis in this indication and extend it to other hospital centers for improve the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* patient who must perform an electromyogram
* patient who have given their free and informed consent

Exclusion Criteria:

* Patient known to be not receptive to hypnosis
* Patient having a contraindication to hypnosis (Psychotic disorders, paranoid personality)
* Patient having cognitive disorders or comprehension problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Quantitative pain | Visual Analog Scale (0 = no pain to 10 = extreme pain) will be completed by the patient 5 minutes before and 5 minutes after the end of the electromyogram
  Evaluation of Pain reduction during the electromyogram following the concomitant practice of hypnosis, assessed quantitatively using the Visual Analog Scale

SECONDARY OUTCOMES:
Qualitative pain | Saint-Antoine Pain Questionary will be completed by the patient 5 minutes before and 5 minutes after the end of the electromyogram
  Evaluation of Pain reduction during the electromyogram following the concomitant practice of hypnosis, assessed qualitatively assessment, using the Saint-Antoine Pain Questionary
Anxiety | Beck Anxiety Inventory (0 = no anxiety to 63 = severe anxiety) will be completed by the patient 5 minutes before and 5 minutes after the end of the electromyogram
  Evaluation of Anxiety assessment using the Beck Anxiety Inventory

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH de Pau, Pau
  - KRIM Elsa, Pau

IPD SHARING:
Plan to Share IPD: Undecided